CLINICAL TRIAL: NCT03786848
Title: A Single-center, Open, Real World and Prospective Trial of Personalized Mini Patient-Derived Xenograft (MiniPDX ) Modeling in Adult Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Personalized Mini-PDX for Metastatic CRPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MiniPDX-CRPC
Record Dates: First submitted 2018-12-06; First posted 2018-12-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Patient Derived Xenograft; CRPC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MiniPDX Group (Experimental): Patients medication plan based on MiniPDX drug sensitivity test.
  Interventions: Other: MiniPDX Group

INTERVENTIONS:
Other: MiniPDX Group — Mini patient derived xenograft (MiniPDX) is a drug sensitivity test model established by transplanting primary human tumor cells into immunodeficient mice by special methods. This test can provide sensitivities of single drug or drug combination within 7 days to screen out the optimal individualized regimens for each patient.

SUMMARY:
The investigators intend to use the Second-generation sequencing（NGS）and MiniPDX drug sensitivity models to guide the treatment decision-making for patients who were resistant to abiraterone, enzalutamide or other new second-generation anti-androgenic drugs. In order to develop precise personalized treatment plans for patients and extent their lifetimes.

DETAILED DESCRIPTION:
Most patients with metastatic prostate cancer are effective in endocrine therapy at the beginning, but after a median survival of 12 to 18 months, almost all patients develop castration-resistant prostate cancer (CRPC). Since the pathogenesis of CRPC is still unknown, the clinical lack of precise treatment for the cause is a difficult and hot topic in current research and treatment. Mini patient derived xenograft (MiniPDX) is a drug sensitivity test model established by transplanting primary human tumor cells into immunodeficient mice by special methods. This efficient drug sensitivity test can provide sensitivities of single drug or drug combination in order to screen out the optimal individualized regimens for each patient. The investigators intend to use the Second-generation sequencing（NGS）and MiniPDX drug sensitivity models to guide the treatment decision-making for patients who were resistant with abiraterone, enzalutamide or other new second-generation anti-androgenic drugs. This project is to develop precise personalized treatment plans for patients and extent their lifetimes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient can provide detailed clinical baseline information including: name, age, gender, pathology, past treatment, etc.;
2. Male, age ≥ 18 years old;
3. ECOG score 0~2 points;
4. Patient must be able to provide tissue samples for the drug sensitive test;
5. No treatment history with PI3K inhibitors, AKT inhibitors or mTOR inhibitors;
6. Estimated lifetime is ≥ 3 months;
7. Histological or cytologically determined prostate adenocarcinoma, excluding neuroendocrine differentiation, signet ring cell carcinoma and small cell carcinoma;
8. Patient is at a castration level and the testosterone level is lower than <50 ng/dL or 1.7 nmol/L;
9. Received abiraterone or enzalutamide and other new second-generation anti-androgenic drugs and have disease progression. Disease progression is defined by PCWG3 :The progression of disease in PCWG3 is defined as satisfying one of the following: according to the increase in PSA levels, there must be three consecutive increases in PSA at least one week apart, and the minimum value is greater than or equal to 5.0 ng/ml; disease progression as assessed by RECIST 1.1, considering PSA levels or not; PCWG3 defines bone disease progression, which is bone scan found 2 or more new lesions;
10. Evidence of distant metastatic disease (such as bone scans and CT/MRI results), imaging data that can be used to assess the condition before and after treatment, or imaging experience provided by three imaging hospitals with experience in three hospitals. Test reports and oncology indicators include PSA values;
11. The patient can tolerate the primary physician to perform the puncture operation, after receiving the informed consent from the patient and the family members;
12. The follow-up period must be at least greater than 2 months;
13. Be able to follow the research and follow-up procedures to provide real and effective information;
14. The patient or his legal guardian understands the test procedure and content and voluntarily signs the printed informed consent form.

Exclusion Criteria:

1. Cognitive ability and psychological abnormalities
2. ECOG score 3-4 points or blood biochemical examination indicates that the patient is not suitable for continuing chemotherapy or chemotherapy has been postponed
3. Can not provide enough tumor puncture tissue, not enough tumor cells for subsequent experiments;
4. Patient who is unwilling to receive follow-up treatment after the Mini PDX model drug sensitivity test;
5. The investigator believes that the subject may not be able to complete the study or may not be able to comply with the requirements of this study (for administrative reasons or other reasons).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-27 (Estimated); Study Completion 2021-01-27 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 months
  The ratio of number of participants with evidence of a confirmed complete response (CR) or partial response (PR) to all participants is objective response rate (ORR) by using Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 to evaluate.

SECONDARY OUTCOMES:
PFS | 12 months
  Progression-free survival (PFS) is defined as the time from the date of the first administration of patients medication plan based on MiniPDX drug sensitivity test to the date of the first documentation of disease progression or death due to any cause, whichever comes first, censored at the last date at which the participant was determined to be progression-free.
OS | 12 months
  Overall survival is defined as time from initiation to death of any cause.
ADR | Up to 30 days of last study treatment.
  Adverse Drug Reaction：Adverse events determined according to CTCAE (version 4.03) and attribution to study treatment.
Clinical Consistency | Up to 2 months of last study treatment.
  Overall clinical consistency（accuracy） as assessed by evaluating Response Evaluation Criteria In Solid Tumors (RECIST) criteria in patient tumor and correlating to tumor regression in Mini-PDX model for same drug treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang F, Wang W, Long Y, Liu H, Cheng J, Guo L, Li R, Meng C, Yu S, Zhao Q, Lu S, Wang L, Wang H, Wen D. Characterization of drug responses of mini patient-derived xenografts in mice for predicting cancer patient clinical therapeutic response. Cancer Commun (Lond). 2018 Sep 26;38(1):60. doi: 10.1186/s40880-018-0329-5. PMID 30257718